CLINICAL TRIAL: NCT05275127
Title: Analysis of Gingival Crevicular Fluid miRNA Changes After Periodontal Treatment.
Brief Title: Impact of Periodontal Treatment on Local miRNA Expression
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Other Study IDs: 215/21/PO
Record Dates: First submitted 2022-02-08; First posted 2022-03-11 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Diseases; Periodontal Diseases
Keywords: Periodontitis, GCF
MeSH Terms: conditions — Cardiovascular Diseases; Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Q-SRP: Evaluation of changes of gingival crevicular fluid miRNA
  Interventions: Other: changes of gingival crevicular fluid miRNA
- FM-SRP: Evaluation of changes of gingival crevicular fluid miRNA
  Interventions: Other: changes of gingival crevicular fluid miRNA

INTERVENTIONS:
Other: changes of gingival crevicular fluid miRNA — Evaluation of changes of gingival crevicular fluid miRNA after periodontal treatment

SUMMARY:
To assess the impact of Fill Mouth Scaling and Root planing or Quadrant Scaling and Root planing gingival crevicular fluid (GCF) levels of miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 100-5p, miRNA 125-5p, miRNA 200b-3p and miRNA 200b-5p and their correlation with periodontitis extent.

DETAILED DESCRIPTION:
The patients selected for the study were divided into 2 groups: group 1 (FM-SRP), group 2 (Q-SRP). Any selected subject underwent anamnestic and periodontal examination, blood and GCF sampling. MiRNA in the GCF was extracted through a commercially available kit and then measured carrying out real-time quantitative polymerase chain reaction (RT-PCR).

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 15 teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL)

  ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Q-SRP (no. 44 patients), FM-SRP (no. 45 patients)
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level reduction | 1-year
  evaluation of millimeters reduction of clinical attachment level (CAL) after periodontal therapy

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — Università degli Studi di Catania
Locations (1):
- University of Catania, Catania, CT, Italy

IPD SHARING:
Plan to Share IPD: Undecided
all collected IPD, all IPD that underlie results in a publication